CLINICAL TRIAL: NCT00088231
Title: Ph I/II Study of PTK 787 (Vatalanib) and Gleevec (Imatinib) in Patients With Refractory Acute Myelogenous Leukemia (AML), Agnogenic Myeloid Metaplasia (AMM), and Chronic Myelogenous Leukemia- Blastic Phase (CML-BP)
Brief Title: PTK 787 and Gleevec in Patients With AML, AMM, and CML-BP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0248
Record Dates: First submitted 2004-07-22; First posted 2004-07-23 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Acute Myelogenous Leukemia; Agnogenic Myeloid Metaplasia; Chronic Myelogenous Leukemia
Keywords: Acute Myelogenous Leukemia (AML); Agnogenic Myeloid Metaplasia (AMM); Chronic Myelogenous Leukemia-Blastic Phase (CML-BP)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — Imatinib Mesylate; vatalanib

ARMS (2):
- PTK 787 + Imatinib (Experimental): For 1 week prior to receipt of study combination regimen, all patients will receive single agent PTK 787 at dose specified for that dose level of the study combination regimen to allow stabilization of PTK 787 levels. Patients should not have a grade 3 or 4 PTK 787-related adverse events in order to begin study combination therapy with a imatinib on day 8. On Day 8, PTK 787 250 mg by mouth every day and imatinib 600 mg by mouth every day (for Acute Myelogenous Leukemia (AML), Chronic Myelogenous Leukemia- blastic phase (CML-BP) and imatinib 400 mg by mouth every day (for Agnogenic Myeloid Metaplasia (AMM). Length of therapy is four courses; each course equals 28 days. Patients assessed for response after each course.
  Interventions: Drug: Imatinib Mesylate (Gleevec); Drug: PTK 787 (vatalanib)
- PTK 787 (vatalanib) Alone (Experimental): For 1 week prior to receipt of study combination regimen, all patients will receive single agent PTK 787 at dose specified for that dose level of the study combination regimen to allow stabilization of PTK 787 levels. Patients should not have a grade 3 or 4 PTK 787-related adverse events in order to begin study combination therapy with a imatinib on day 8. PTK 787 250 mg by mouth for Days 1 - 7.
  Interventions: Drug: PTK 787 (vatalanib)

INTERVENTIONS:
Drug: Imatinib Mesylate (Gleevec) — 600 mg by mouth every day (for AML, CML-BP) for a 28 day cycle.
  400 mg by mouth every day (for AMM) for a 28 day cycle.
  Other Names: Imatinib; Gleevec; ST1571; NSC-716051
  Arms: PTK 787 + Imatinib
Drug: PTK 787 (vatalanib) — For 1 week prior to receipt of the study combination regimen, all patients will receive single agent PTK 787 at the dose specified for that dose level of the study combination regimen to allow stabilization of PTK 787 levels.
  Starting dose: 250 mg by mouth every day for a 28 day cycle.
  Other Names: Vatalanib

SUMMARY:
The goal of this clinical research study is to find the highest safe doses of PTK 787 (vatalanib) and Gleevec (imatinib mesylate) that can be given to treat Chronic Myelogenous Leukemia-Blastic Phase (CML-BP), Refractory Acute Myelogenous Leukemia (AML), or Agnogenic Myeloid Metaplasia (AMM). Another goal is to see how effective this combination treatment is.

DETAILED DESCRIPTION:
Rationale: The purpose of this study is to combine PTK-787, a potent orally vascular endothelial growth factor (VEGF) receptor inhibitor (in disorders where VEGF is known to be involved in the pathophysiology), with Imatinib mesylate (IM), a protein-tyrosine kinase inhibitor of abl, Bcr-Abl, platelet derived growth factor (PDGF), and c-Kit (in same disorders where these kinases are believed to be important). The potential synergy between oral agents that inhibit these kinases in disorders where each of the two agents have some, but inadequate, single agent activity is being studied in this protocol. We will also have an opportunity to assess if there is any correlation between response and individual kinase mutations e.g., c-Kit in patients with AML. If improved outcomes are observed, further studies will be indicated to investigate which, if either, agent is predominantly responsible for such a benefit - these studies will be facilitated by the availability of more potent e.g., (AMN107 as an abl inhibitor), (Bevacizumab, AG013736 as VEGF inhibitors) agents which will help to define the relative importance of the various inhibitory activities.

Objectives: To determine the maximum tolerated doses (MTD) and pharmacokinetics (PK) of PTK 787 and imatinib mesylate, when given in combination to patients with refractory acute myelogenous leukemia (AML), agnogenic myeloid metaplasia (AMM) and chronic myelogenous leukemia in blastic phase (CML-BP).

To determine the efficacy (response rate, survival, time to progression, time to treatment failure, duration of response) of the MTD in these study populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML (including refractory anemia with excess of blasts [RAEB], refractory anemia with excess of blasts in transition to AML [RAEBT], or untreated AML when standard chemotherapy is not considered appropriate or is refused, CML in blastic phase, and agnogenic myeloid metaplasia (AMM)
* Age 15 years or greater (separate pediatric studies will be conducted if results of adult studies are considered sufficiently positive)
* Laboratory values less than or equal to 2 weeks prior to study entry - Serum bilirubin 1.5mg/dL, unless considered due to organ leukemic involvement or Gilbert's syndrome. - SGOT or SGPT less than or equal to 2.5 x upper limit of normal. - Serum creatinine less than or equal to 2mg/dL,
* Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein less than or equal to 500 mg and measured creatinine clearance (CrCl) greater than or equal to 50 mL/min from a 24-hour urine collection.
* The effects of PTK 787 and imatinib on the developing human fetus are unknown. For this reason and because inhibitors of mRNA translation are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) for the duration of study participation.
* Due to possible interactions with study drugs, oral contraceptives should not be used. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. If the partner of a male patient taking PTK 787 and/or Gleevec conceives, the physician should be notified
* Ability to understand and the willingness to sign a written informed consent document.
* Performance Status less than or equal to 2.

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy, except for hydroxyurea, or radiotherapy within 7 days prior to entering the study. Patients will have cleared all toxicities from prior therapies before starting this study combination.
* Patients who have received investigational drugs less than or equal to 2 weeks prior to study entry
* Prior therapy with anti-VEGF agents.
* Concomitant administration of anticancer drugs is not permitted, except for hydroxyurea. Leukopheresis is allowed within the first 28 days of treatment if required to control elevated blast levels or platelet counts. Within the first 28 days of treatment, hydroxyurea may be given at a maximum dose of 5 g daily for up to a total of 7 days. For leukopheresis, a maximum of 2 procedures per week or 4 procedures during the first 28 days is allowed.
* Patients may not be receiving any other cytotoxic investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PTK 787 or imatinib.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled diabetes, interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung, chronic liver disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Uncontrolled intercurrent illness including, not limited to, ongoing uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled high blood pressure, history of labile hypertension, history of poor compliance with an antihypertensive regimen, myocardial infarction less than or equal to 6 months prior to registration, uncontrolled diabetes, interstitial pneumonia or extensive and symptomatic interstitial fibrosis of lung, chronic liver disease or psychiatric illness/social situations that limits compliance with study requirements.
* Pleural effusion or ascites that causes respiratory compromise (greater than or equal to Common Toxicity Criteria (CTC) grade 2 dyspnea).
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets).
* Patients with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded - A separate study for patients with HIV will be performed if indicated.
* Pregnant women are excluded from this study because PTK 787 and imatinib may have a potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PTK 787 or imatinib, breastfeeding patients will not be eligible.
* Patients with known central nervous system (CNS) disease are excluded.
* Patients with a history of another primary malignancy less than or equal to 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin.
* Patients w/ recent major surgery are excluded (less than 4 wks of starting this study) or minor surgery less than or equal to 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities.
* Patients who are taking warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin is allowed.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Time to Response | 28 days
  Time to response is defined as the period of time from the date of first study drug administration until the first objective documentation of response.

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org